CLINICAL TRIAL: NCT03292146
Title: Effects of Denosumab on Bone Mineral Density, Markers of Bone Metabolism and Bone Microarchitecture in Women With Anorexia Nervosa: A Pilot Study
Brief Title: Effects of Denosumab on Bone Mineral Density in Women With Anorexia Nervosa: A Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P000529
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2022-09

CONDITIONS: Bone Density; Bone Loss; Anorexia Nervosa; Eating Disorder; Atypical Anorexia Nervosa
MeSH Terms: conditions — Bone Diseases, Metabolic; Anorexia Nervosa; Feeding and Eating Disorders | interventions — Denosumab; Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Denosumab 60mg Injection (Experimental): Denosumab 60mg injection at baseline study visit and 6 month study visit. Alendronate 70mg PO weekly starting at Month 12 through 24 months.
  Interventions: Drug: Denosumab 60 MG [Prolia]; Drug: Alendronate 70Mg Tab
- Placebo (Placebo Comparator): Placebo injection at baseline study visit and 6 month study visit. Alendronate 70mg PO weekly starting at Month 12 through 24 months.
  Interventions: Drug: Placebo Injection; Drug: Alendronate 70Mg Tab

INTERVENTIONS:
Drug: Denosumab 60 MG [Prolia] — Denosumab 60mg injection at baseline and 6 months
  Arms: Active Denosumab 60mg Injection
Drug: Placebo Injection — Placebo Injection at baseline and 6 months
  Arms: Placebo
Drug: Alendronate 70Mg Tab — Alendronate 70mg PO weekly starting at Month 12 through 24 months.

SUMMARY:
This protocol is a randomized, double-blind, placebo-controlled clinical trial which aims to investigate the effect of denosumab on BMD in women with anorexia nervosa. The investigators hypothesize that 12 months of denosumab administration will result in an increase in bone mineral density, decrease in markers of bone resorption and improvement in bone microarchitecture in osteopenic women with anorexia nervosa compared with placebo.

An optional extension study will offer subjects 12-month administration of open-label alendronate (an oral bisphosphonate) after the initial 12 month administration of denosumab or placebo. We hypothesize that 12 months of denosumab followed by 12 months of open-label alendronate will result in a greater increase in BMD compared to 12 months of placebo followed by 12 months of open-label alendronate. Within the group of women who receive sequential therapy with 12 months of denosumab followed by 12 months of alendronate, we hypothesize that BMD will be maintained between 12 and 24 months while on alendronate.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Inclusion Criteria:

* Female
* Age 20-60 years, skeletally mature with closed epiphyses
* Anorexia nervosa or atypical anorexia nervosa defined by DSM-V diagnostic criteria
* BMD T-score < -1.0
* Normal serum 25-OH vitamin D (>30 ng/mL) and calcium levels
* For women of reproductive age, agree to use an effective contraceptive method. Highly effective methods of birth control include:

  * Combined (estrogen and progestogen) hormonal methods (pills, vaginal ring, or skin patch)
  * Intrauterine device (IUD)
  * Intraduterine hormonal-releasing system (IUS)
  * Surgery to tie both fallopian tubes (bilateral tubal ligation/occlusion)
  * Your male partner has had a vasectomy and testing shows there is no sperm in the semen
* Dental check up within the past year

Exclusion Criteria:

* Any disease known to affect bone, including untreated thyroid dysfunction, Cushing's or renal failure
* Subjects with a known esophageal disease cannot participate in the alendronate extension study
* Any medication known to affect bone metabolism within 3 months of the study, excluding oral contraceptives or other forms of estrogen administration. Bisphosphonates must have been discontinued for at least one year before participation
* Immunodeficiency or taking immunosuppressive therapy
* Serum potassium <3.0 meq/L
* Serum ALT >3 times upper limit of normal
* eGFR of less than 30 ml/min
* Hypocalcemia
* Diabetes mellitus
* Active substance abuse, including alcohol
* History of malignancy
* Paget disease of bone
* Osteomalacia
* Osteonecrosis of the jaw (ONJ) or risk factor for ONJ, such as invasive dental procedures (eg, tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal and/or pre-existing dental disease, and current use of corticosteroids.
* Planned invasive dental procedure over the next 24 months.
* Known senstivity to any of the products or components to be administered during dosing or known sensitivity to mammalian cell derived drug products
* Sensitivity to calcium or vitamin D supplements
* Pregnant, planning to become pregnant with 7 months after the end of treatment and/or breastfeeding

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women, age 20-60 years, with anorexia nervosa or atypical anorexia nervosa and BMD T-score < -1.0
Pre-assignment Details: Randomized, double-blind, placebo-controlled trial. 30 subjects randomized in a 2:1 ratio to denosumab followed by alendronate or placebo followed by alendronate groups
Groups:
- Denosumab (0-12 months) followed by alendronate (12-24 months): Denosumab 60 mg SQ injections q6 months for 12 months followed by alendronate 70 mg PO weekly for 12 months.
- Placebo (0-12 months) followed by alendronate (12-24 months): Placebo SQ injections q6 months for 12 months followed by alendronate 70 mg PO weekly for 12 months.
Period: Baseline to 12 months
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
Started | 20 | 10
Completed | 18 | 9
Not Completed | 2 | 1
Not completed — Relocation | 1 | 0
Not completed — Seeking higher level of care for eating disorder | 1 | 0
Not completed — Seeking treatment for chronic fatigue syndrome | 0 | 1
Period: 12 months to 24 months
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
Started | 18 | 9
Completed | 15 | 6
Not Completed | 3 | 3
Not completed — Planning pregnancy | 2 | 2
Not completed — Personal reasons | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Women, age 20-60 years, with anorexia nervosa or atypical anorexia nervosa and BMD T-score < -1.0
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months) | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (8.0) | 29.4 (6.8) | 29.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 10 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
Body mass index (BMI) [Mean (Standard Deviation); unit: kg / m^2] | 19.0 (1.7) | 18.0 (2.0) | 18.7 (1.9)
Postero-anterior (PA) lumbar spine areal bone mineral density (aBMD) Z-score [Mean (Standard Deviation); unit: Z-score] — PA lumbar spine aBMD Z-score was obtained by dual-energy x-ray absorptiometry (DXA). A BMD Z-score is the number of standard deviations above or below the mean BMD given a person's age, sex, and race. A BMD Z-score of "0" represents the population mean. A BMD Z-score >0 represents a higher/better BMD, whereas a BMD Z-score <0 represents a lower/worse BMD. A BMD Z-score between -1 and -2.5 signifies osteopenia. A BMD Z-score at or below -2.5 signifies osteoporosis.
  Z-score | -1.6 (0.9) | -1.7 (1.4) | -1.6 (1.1)
Postero-anterior (PA) lumbar spine aBMD [Mean (Standard Deviation); unit: g/cm^2] | 0.86 (0.09) | 0.85 (0.16) | 0.86 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Postero-anterior (PA) Lumbar Spine Bone Mineral Density by Dual-energy X-ray Absorptiometry (DXA)
Description: Postero-anterior (PA) lumbar spine bone mineral density was assessed by dual-energy x-ray absorptiometry (DXA). The DXA scanner used was a Hologic Horizon A (Hologic, Inc., Waltham, MA).
Time Frame: 12 months (Period 1)
Population: Women, age 20-60 years, with anorexia nervosa or atypical anorexia nervosa and BMD T-score < -1.0
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
Number analyzed (Participants) | 20 | 10
g/cm^2 | 0.90 (0.03) | 0.87 (0.04)
Statistical Analysis 1: Comparison: Denosumab (0-12 months) followed by alendronate (12-24 months) vs Placebo (0-12 months) followed by alendronate (12-24 months); Test type: Superiority; p = 0.009, Mixed Models Analysis

2. Secondary Outcome: Percent Change Postero-anterior (PA) Lumbar Spine Bone Mineral Density by DXA
Time Frame: Baseline to 24 months
Population: Women ages 20-60 with anorexia nervosa/atypical anorexia nervosa and BMD T-score < -1.0
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
Number analyzed (Participants) | 20 | 10
% change | 3.9 (4.3) | 5.8 (5.3)
Statistical Analysis 1: Comparison: Denosumab (0-12 months) followed by alendronate (12-24 months) vs Placebo (0-12 months) followed by alendronate (12-24 months); Test type: Superiority; p = 0.41, t-test, 2 sided

3. Secondary Outcome: Percent Change Postero-anterior (PA) Lumbar Spine Bone Mineral Density by DXA
Time Frame: 12 months to 24 months (Period 2)
Population: Women ages 20-60 with anorexia nervosa/atypical anorexia nervosa and BMD T-score < -1.0
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
Number analyzed (Participants) | 20 | 10
% change | -2.0 (3.7) | 4.6 (3.2)
Statistical Analysis 1: Comparison: Denosumab (0-12 months) followed by alendronate (12-24 months); Test type: Superiority; p = 0.06, Matched pairs
Statistical Analysis 2: Comparison: Placebo (0-12 months) followed by alendronate (12-24 months); Test type: Superiority; p = 0.01, Matched pairs

ADVERSE EVENTS:
Time Frame: Baseline to 24 months
Description: Serious adverse events reported to the IRB immediately upon the PI becoming aware.
Arm/Group | Denosumab (0-12 months) followed by alendronate (12-24 months) | Placebo (0-12 months) followed by alendronate (12-24 months)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 6/20 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denosumab (0-12 months) followed by alendronate (12-24 months) (N=20) | Placebo (0-12 months) followed by alendronate (12-24 months) (N=10)
constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
nausea/stomach pain/bloating (Gastrointestinal disorders) | 1 (2) | 0 (0)
bone fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Unrelated injury
Keratitis (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder biliary dyskinesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
C. difficile (Infections and infestations) | 1 (1) | 0 (0)
Disc degeneration and herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03292146/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03292146/SAP_001.pdf